CLINICAL TRIAL: NCT06390774
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of SSGJ-705 Monotherapy in Patients with Advanced Malignant Tumors
Brief Title: A Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of SSGJ-705 Monotherapy in Patients with Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-705-CA-Ⅰ-01
Record Dates: First submitted 2024-04-08; First posted 2024-04-30 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Locally Advanced, Recurrent or Metastatic Malignancies
Keywords: advanced malignancies
MeSH Terms: conditions — Recurrence; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1 (Experimental): Dose escalation will be conducted using a traditional 3+3 design. Dose Escalation includes 6 levels, QW IV. Dose extension will be carried out at the selected level.
  Interventions: Drug: SSGJ-705
- Part 2 (Experimental): Dose escalation will be conducted using a traditional 3+3 design. Dose Escalation includes 6 levels, Q2W IV. Dose extension will be carried out at the selected level.
  Interventions: Drug: SSGJ-705
- Part 3 (Experimental): Dose escalation will be conducted using a traditional 3+3 design. Dose Escalation includes 6 levels, Q3W IV. Dose extension will be carried out at the selected level.
  Interventions: Drug: SSGJ-705
- Part 4 (Experimental): Indication extension will be carried out at the selected level，including 3 dosage levels.
  Interventions: Drug: SSGJ-705

INTERVENTIONS:
Drug: SSGJ-705 — anti-PD-1 and anti-HER2 bispecific antibody

SUMMARY:
This study was an open-label phase I study to evaluate the safety, tolerability, PK profile and potential efficacy of SSGJ-705 as a single agent in patients with advanced malignancies.

DETAILED DESCRIPTION:
This study includes 4 Parts: Part 1 (dose escalation and dose extension for QW administration), Part 2 (dose escalation and dose extension for Q2W administration), Part 3 (dose escalation and dose extension for Q3W administration), and Part 4 (indication extension, such as HER2 expression, PD-L1 high expression, driver gene negative newly treated advanced NSCLC, or other tumors).

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females over age 18
2. Histologically and/or cytologically documented local advanced or recurrent or metastatic malignancies
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Expected survival >3 months.
5. Signed informed consent form.
6. Must have adequate organ function.

Exclusion Criteria:

1. Any remaining AEs > grade 1 from prior anti-tumor treatment as per CTCAE v5. 0, with exception of hair loss, fatigue, and grade 2 peripheral neurotoxicity.
2. Pregnant or nursing women or women/men who are ready to give birth
3. Symptomatic central nervous system metastasis.
4. Allergy to other antibody drugs or any excipients in the study drugs.
5. Severe dyspnea at rest due to complications of advanced malignant tumors, or needing supplemental oxygen therapy.
6. Participated in any clinical study of medical devices or drugs within 1 month prior to screening (excluding non-intervention clinical studies or follow-up period of intervention clinical studies) .

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
DLTs | 14 days
  Dose limiting toxicity
AE | up to 1 year
  Safety and tolerability assessed by incidence and severity of adverse events
MTD or MAD | up to 1 year
  maximum tolerated dose or the maximum administered dose if MTD is not reached
RP2D | up to 1 year
  the recommended phase II dose

SECONDARY OUTCOMES:
ORR | up to 1 year
  Objective response rate
PFS | up to 1 year
  Progression-free Survival
Cmax | up to 1 year
  Maximum Plasma Concentration
T1/2 | up to 1 year
  Half-life

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Cancer Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No